CLINICAL TRIAL: NCT02427113
Title: What Are the Effects of Music on TMD Symptoms?
Brief Title: What Are the Effects of Music on Temporomandibular Disorder Symptoms?
Acronym: TMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Alicia Howard, PhD Candidate, University of Toronto, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZurichUAS
Record Dates: First submitted 2015-03-25; First posted 2015-04-27 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: TMD
Keywords: TMD; Music Medicine; Vibroacousitc Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Select Music (Active Comparator): Participants will be randomized to two groups. Self-select music will be used as treatment for managing pain. They will be required to listen to their preferred songs for 30 minutes per 7 days, recommended 5, for 3 weeks.
  Interventions: Other: Self-Select Music
- Sound Oasis Vibrating Chair (Active Comparator): Participants will be randomized to two groups. Vibroacoustic therapy will be administered in the form of a vibrating chair. They will be required to listen to their preferred songs for 30 minutes per 7 days, recommended 5, for 3 weeks.
  Interventions: Other: Sound Oasis Vibrating Chair

INTERVENTIONS:
Other: Sound Oasis Vibrating Chair — Sound oasis vibroacoustic chair will be used as treatment for managing TMD related pain
  Arms: Sound Oasis Vibrating Chair
Other: Self-Select Music — The self-select music of the participants will be applied for managing the painful symptoms of TMD
  Arms: Self-Select Music

SUMMARY:
The purpose of the study will be to examine the effectiveness of an innovative use of music on TMD. Music and rhythmic vibrations can alter the basic processes related to sensation of pain in the brain. As well, music can block the neurological pathways that transmit pain sensations and thereby reduce pain. Music and vibrations are relaxing, reduce stress, and thereby reduce sensitivity to pain.

DETAILED DESCRIPTION:
The investigators hypothesize that patients will experience less pain, an elevation in mood, a decrease in stress, higher well-being, and a reduction in TMD symptoms after receiving therapeutic music treatments. The investigators further predict that the vibrations generated by the Sound Oasis VTS1000 (vibroacoustic chair) will produce stronger effects than self-selected music. The question to be investigated in this study: "What are the effects of music on TMD symptoms?"

Participant intake will occur prior to study providing information on diagnostics, music preferences, participant demographics, and participant randomization. The study will consist of 4 assessments and 2 treatments with a 1 month wash-out period between treatments. Assessment 1 (will serve as pre-test) and occur before 1st treatment. Assessment 2 (will serve as post-test), taking place before 2nd treatment and will last 45 minutes. Assessment 3 will follow the wash-out period; and assessment 4 (the final session), which will be a total of 60 minutes will include a participant treatment review interview. Pre/post assessments will be utilized as a means to examine change in pain at the level of each participant, mood levels, depression and the perception of quality of life.

Therapeutic music treatments, which will consist of randomly assigned interventions of Sound Oasis VTS-1000 and preferred music playlist, will be prescribed for self-administered in-home sessions for 3-weeks, 7 days (recommended) but at least a minimum of 5 days per week. During each 3-week music treatment period, 1 self-administered in-home music treatment will be prescribed for 3-weeks, 7 days (recommended) but at least a minimum of 5 days per week.

There will be 2 times where the participants receive no therapeutic music intervention but will continue with treatment as usual which will occur 7 days prior to each treatment. Participants will be asked to do a daily pain rating for one week during treatment as usual before the start of the music interventions.

There will be a 4-week wash-out period between therapeutic music treatments 1 and 2. There will be no music treatment during this time. Participants will be asked to keep a record of the type of medication taken, a pill count, and frequency of medication during this time as well as during treatment.

Both therapeutic music and treatment as usual times will be intervened by a treatment compliance email or phone call by the music therapist. Participants will be randomly assigned to 2 groups: (a) Sound Oasis VTS-1000 and (b) participant preferred music. Participants will complete questionnaires at the beginning of the study, following the end of the first 3 weeks of either therapeutic music treatment, at the end of the second 3 weeks of therapeutic music and during the final assessment time, which will also consist of a brief interview about treatment received.

Data will be analyzed with reference given only to an assigned ID number. All information collected will be used for this study to investigate the effects of therapeutic music on the management of TMD symptoms. Furthermore, all participants will be informed that all information that will be disclosed will remain confidential, unless the disclosed information will cause harm to self or others.

ELIGIBILITY:
Inclusion Criteria:

* hearing able as listening to music is required as part of treatment
* main source of pain is myofascial pain
* on-going pain for 6 months

Exclusion Criteria:

* Acute Inflammatory Conditions - an inflammation having a rapid onset, with a clear and distinct termination. (e.g. Rheumatoid arthritis and Osteoarthritis)
* Clients Presenting with Psychoses
* Pregnancy
* Hemorrhaging or Active Bleeding
* Thrombosis
* Hypotension
* Pacemakers as contraindications of Vibroacoustic Therapy (VAT) are related to these conditions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale to measure pain levels | 3 months
  A psychometric response scale which can be used in questionnaires to measure participants pain levels.

SECONDARY OUTCOMES:
Short Inventory Depression Scale | 3 months

OTHER OUTCOMES:
Mult-Dimensional Mood Questionnaire | 3 months
Quality of Life Enjoyment and Satisfaction Questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Allan Gordon, PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital's Wasser Pain Management Centre, Toronto, Ontario, Canada